CLINICAL TRIAL: NCT00712582
Title: Risk-Adapted Therapy for Patients With Untreated Age-Adjusted International Prognostic Index Low-Intermediate Risk, High-Intermediate Risk, or High Risk Diffuse Large B Cell Lymphoma
Brief Title: Therapy for Patients With Untreated Age-Adjusted International Prognostic Index Low-Intermediate Risk, High-Intermediate Risk, or High Risk Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-026
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2021-03

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin; Lymphoma; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; ifosfamide; etoposide; carboplatin; stem cell transplant; 08-026
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Etoposide; Carboplatin; Ifosfamide; Rituximab; Mitoxantrone; Cyclophosphamide; Carmustine

ARMS (3):
- Consolidation A (Experimental): Induction: RR-CHOP-14 Chemotherapy for Three Cycles Each cycle lasts approximately 14 days. A total of 3 cycles of RR-CHOP-14 will be given. One cycle of CHOP will follow.
  Patients whose disease is FDG-PET negative or patients whose FDG-PET scan is positive but repeat biopsy is negative and whose initial Ki-67 expression is < 80% will receive 3 cycles of standard dose ICE Chemotherapy.
  Interventions: Drug: Etoposide, carboplatin, ifosfamide
- Consolidation B (Experimental): Induction: RR-CHOP-14 Chemotherapy for Three Cycles Each cycle lasts approximately 14 days. A total of 3 cycles of RR-CHOP-14 will be given. One cycle of CHOP will follow.
  Patients whose disease is FDG-PET negative or patients whose FDG-PET scan is positive but repeat biopsy is negative and whose initial Ki-67 expression is ≥80% will receive 2 cycles of augmented RICE Chemotherapy (as per MSKCC protocol 03-075).
  Interventions: Drug: Rituximab, Ifosfamide, Etoposide, Carboplatin
- Consolidation C (Experimental): Induction: RR-CHOP-14 Chemotherapy for Three Cycles Each cycle lasts approximately 14 days. A total of 3 cycles of RR-CHOP-14 will be given. One cycle of CHOP will follow.
  Consolidation C: Patients with biopsy proven disease after induction therapy. Patients whose bone marrow remain positive at interim restaging will have the option of getting an allogeneic[m3] stem cell transplant, in lieu of an ASCT, if they have an acceptable HLA match donor. The allogeneic[m4] stem cell transplant regimen will be decided by the MSK Bone Marrow Transplant Service.
  Interventions: Drug: Rituximab, Ifosfamide, Etoposide, Carboplatin, Stem Cell Collection, Mitoxantrone, Cyclophosphamide and etoposide, Carmustine

INTERVENTIONS:
Drug: Etoposide, carboplatin, ifosfamide — Patients in consolidation A will receive three drugs in a regimen called ICE. You will have 3 cycles. Each new cycle begins 2 to 3 weeks after the last one.
  Arms: Consolidation A
Drug: Rituximab, Ifosfamide, Etoposide, Carboplatin — It consists of four drugs in a regimen called augmented RICE (augRICE). It is given every 3 weeks for 2 cycles.
  Arms: Consolidation B
Drug: Rituximab, Ifosfamide, Etoposide, Carboplatin, Stem Cell Collection, Mitoxantrone, Cyclophosphamide and etoposide, Carmustine — It consists of four drugs in a regimen called augRICE. It is given every 3 weeks for 2 cycles. After the rituximab on day 3, you will then be admitted to the hospital for 2 to 3 nights.
  Part 2: Stem Cell Collection, Part 3: High dose chemoradiotherapy and stem cell transplant. Your doctor may want you to get radiation therapy. If so, it will start 2 weeks before the highdose chemotherapy. This regimen is called CBV-N chemotherapy. It is given by vein in the hospital.
  Arms: Consolidation C

SUMMARY:
About 60% of patients with DLBCL can be cured with a chemotherapy program. It is called RCHOP-21 (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone). It is given once every 3 weeks, for 18 weeks. Each three weeks is a cycle. Some factors predict that you may not be cured with R-CHOP-21. The most common ones are:

* Stage - how much DLBCL, PMBL, or FL3B you have
* LDH - a blood chemistry marker; and
* Whether you can do your normal daily activities. (performance status) We think that the best way to cure more patients with poor risk factors is to add new treatment to R-CHOP. You will get different chemotherapy after 4 cycles. This type of treatment is called risk-adapted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of diffuse large B cell lymphoma, PMLBL, or follicular lymphoma grade 3B confirmed by the department of hematopathology at MSKCC: Patients with discordant bone marrow involvement (i.e. involvement by small cleaved cells or small lymphocytic lymphoma) are eligible.
* Tumors express CD20 as determined by immunohistochemistry.

  o Ki-67 evaluation of tumor tissue
* Patients must have stage III, or IV disease. Patients with IIX, disease must have at least one other age-adjusted IPI risk factor.

  * KPS ≤ 70
  * LDH > upper limit of normal
* All patients must have FDG-PET avid (minimum SUV 2.5) measurable disease
* Patients must have normal baseline cardiac function based upon echocardiogram or gated blood pool scan (MUGA) with an ejection fraction ≥ 50%
* Patients must have a serum creatinine of ≤ 1.5 mg/dl; if creatinine >1.5 mg/dl creatinine clearance must be >60 ml/minute.
* Patients must have ANC>1000/mcl and Platelets>50,000/mcl. If patient has cytopenias due to bone marrow involvement, these requirements are not applicable.
* Patients must have a bilirubin level of < 2.0 mg/dl in the absence of a history of Gilbert's disease (or pattern consistent with Gilbert's)
* Patients must be Hepatitis B surface antigen negative, Hepatitis B core antibody negative, and Hepatitis C negative.
* All patients of childbearing and child creating age must be using an acceptable form of birth control from the initiation of treatment on study until 1 year after completion of chemotherapy and/or transplant.
* Women who are pre-menopausal must have a negative pregnancy test
* Age between 18 and 65
* Patients must be HIV negative. This test may be pending in a patient without risk factors, as determined by the patient's physician.
* If patients have a history of malignancy other than cutaneous basal cell or squamous cell carcinoma, they must be disease-free for ≥ 5 years at the time of enrollment.
* Patients or their guardians must be capable of providing informed consent.
* Patients must be suitable to undergo stem cell transplant.

Exclusion Criteria:

* Any lymphoma subtype other than DLBCL, PMLBL, follicular lymphoma grade 3B
* Patients with either parenchymal brain or lepto-meningeal involvement.
* No more than 14 days of prednisone therapy between the diagnostic biopsy of either DLBCL, PMLBL, or follicular lymphoma grade 3B and the initiation of treatment on study.
* Known pregnancy or breast-feeding
* Medical illness unrelated to NHL which in the opinion of the attending physician and principal investigator will preclude administration of chemotherapy safely. This includes patients with uncontrolled infection, chronic renal insufficiency, myocardial infarction within the past 6 months, unstable angina, cardiac arrhythmias other than chronic atrial fibrillation and chronic active or persistent hepatitis, or New York Heart Association Classification III or IV heart disease.
* History of any malignancy for which the disease-free interval is <5 years, excluding curatively treated cutaneous basal cell or squamous cell carcinoma and carcinoma in-situ of the cervix.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zelenetz, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Bantilan KS, Smith AN, Maurer MJ, Teruya-Feldstein J, Matasar MJ, Moskowitz AJ, Straus DJ, Noy A, Palomba ML, Horwitz SM, Hamlin PA, Portlock CS, Cerhan JR, Habermann TM, Salles GA, Nowakowski GS, Moskowitz CH, Zelenetz AD. Matched control analysis suggests that R-CHOP followed by (R)-ICE may improve outcome in non-GCB DLBCL compared with R-CHOP. Blood Adv. 2024 May 14;8(9):2172-2181. doi: 10.1182/bloodadvances.2023011408. PMID 38271621
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Consolidation A: Induction: RR-CHOP-14 Chemotherapy for Three Cycles Each cycle lasts approximately 14 days. A total of 3 cycles of RR-CHOP-14 will be given. One cycle of CHOP will follow.
  Patients whose disease is FDG-PET negative or patients whose FDG-PET scan is positive but repeat biopsy is negative and whose initial Ki-67 expression is < 80% will receive 3 cycles of standard dose ICE Chemotherapy.
  Etoposide, carboplatin, ifosfamide: Patients in consolidation A will receive three drugs in a regimen called ICE. You will have 3 cycles. Each new cycle begins 2 to 3 weeks after the last one.
- Consolidation B: Induction: RR-CHOP-14 Chemotherapy for Three Cycles Each cycle lasts approximately 14 days. A total of 3 cycles of RR-CHOP-14 will be given. One cycle of CHOP will follow.
  Patients whose disease is FDG-PET negative or patients whose FDG-PET scan is positive but repeat biopsy is negative and whose initial Ki-67 expression is ≥80% will receive 2 cycles of augmented RICE Chemotherapy (as per MSKCC protocol 03-075).
  Rituximab, Ifosfamide, Etoposide, Carboplatin: It consists of four drugs in a regimen called augmented RICE (augRICE). It is given every 3 weeks for 2 cycles.
- Consolidation C: Induction: RR-CHOP-14 Chemotherapy for Three Cycles Each cycle lasts approximately 14 days. A total of 3 cycles of RR-CHOP-14 will be given. One cycle of CHOP will follow.
  Consolidation C: Patients with biopsy proven disease after induction therapy. Patients whose bone marrow remain positive at interim restaging will have the option of getting an allogeneic[m3] stem cell transplant, in lieu of an ASCT, if they have an acceptable HLA match donor. The allogeneic[m4] stem cell transplant regimen will be decided by the MSK Bone Marrow Transplant Service.
  Rituximab, Ifosfamide, Etoposide, Carboplatin, Stem Cell Collection, Mitoxantrone, Cyclophosphamide and etoposide, Carmustine: It consists of four drugs in a regimen called augRICE. It is given every 3 weeks for 2 cycles. After the rituximab on day 3, you will then be admitted to the hospital for 2 to 3 nights.
  Part 2: Stem Cell Collection, Part 3: High dose chemoradiotherapy and stem cell transplant. Your doctor may want you to get radiation therapy. If so, it will start 2 weeks before the highdose chemotherapy. This regimen is called CBV-N chemotherapy. It is given by vein in the hospital.
Period: Overall Study
Arm/Group | Consolidation A | Consolidation B | Consolidation C
Started | 60 | 32 | 4
Completed | 60 | 32 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Consolidation A | Consolidation B | Consolidation C | Total
Number analyzed (Participants) | 60 | 32 | 4 | 96
Age, Continuous [Median (Full Range); unit: years] | 52 [21 to 71] | 49.5 [21 to 69] | 59 [55 to 68] | 51.45 [21 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 19 | 1 | 49
  Male | 31 | 13 | 3 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 60 | 32 | 4 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 60 | 32 | 4 | 96
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 32 | 4 | 96

OUTCOME MEASURES:

1. Primary Outcome: 2-year PFS From the Start of Induction Therapy Conditional
Description: 2-year PFS from the start of induction therapy conditional on attaining either a negative FDG-PET or a negative biopsy at the interim evaluation.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Consolidation A | Consolidation B | Consolidation C
Number analyzed (Participants) | 60 | 32 | 4
percentage of patients | 86.6 [78.4 to 95.7] | 90.6 [81.1 to 100.0] | 0.4 [0.2 to 0.5]

2. Secondary Outcome: Overall Survival at 1 Year
Description: Overall survival from the start of induction therapy conditional on attaining either a negative FDG-PET or a negative biopsy at the interim evaluation.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Percent of patients
Arm/Group | Consolidation A | Consolidation B | Consolidation C
Number analyzed (Participants) | 60 | 32 | 4
Percent of patients | 98.3 [95.1 to 100.0] | 96.9 [91.0 to 100.0] | 50.0 [18.8 to 100.0]

3. Secondary Outcome: Proliferation Marker [18F] Fluorothymidine (FLT) is Significantly Predictive of Progression Free Survival/PFS Via a Log Rank Test.
Description: Obtain preliminary data on potential clinical usefulness of the proliferation marker [18F] fluorothymidine (FLT) in pts with diffuse large cell lymphoma, using combined (FDG-PET/CT). 18F-FLT uptake by visual analysis (stratified as grades 1-3 vs grades 4-5)
Time Frame: Through study completion, up to 10 years
Population: N/A - data were not collected
Arm/Group | Consolidation A
Number analyzed (Participants) | 0

4. Secondary Outcome: Proliferation Marker [18F] Fluorothymidine (FLT) Significantly Predictive of Overall Survival/OS Via a Log Rank Test.
Description: as for outcome 3
Time Frame: Through the completion of study, up to 10 years
Population: N/A - data were not collected
Arm/Group | Consolidation A
Number analyzed (Participants) | 0

5. Secondary Outcome: To Determine the Role of CT Volumetric Analysis Compared to Standard Unidimensional CT in This Patient Population.
Time Frame: conclusion of study
Population: N/A - Data were not collected
Arm/Group | Consolidation A | Consolidation B | Consolidation C
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Consolidation A | Consolidation B | Consolidation C
All-Cause Mortality (participants affected / at risk) | 5/60 | 1/32 | 2/4
Serious Adverse Events (participants affected / at risk) | 15/60 | 12/32 | 2/4
Other Adverse Events (participants affected / at risk) | 0/60 | 0/32 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Consolidation A (N=60) | Consolidation B (N=32) | Consolidation C (N=4)
Allerg react/hypersens (incl drug fever) (Immune system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Blood/Bone Marrow, other (Blood and lymphatic system disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Creatinine (Investigations) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 8 | 0
Fever (in the absence of neutropenia) (General disorders) | 2 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 3 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Leukocytes (Investigations) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1
Neutrophils/granulocytes (Investigations) | 0 | 1 | 0
Pain - Anus (Gastrointestinal disorders) | 0 | 1 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain - Chest/thorax NOS (General disorders) | 0 | 0 | 2
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain - Rectum (Gastrointestinal disorders) | 1 | 0 | 0
Phlebitis (incl superficial thrombosis) (Vascular disorders) | 1 | 1 | 0
Platelets (Investigations) | 3 | 1 | 0
Pneumonia (lung) (Infections and infestations) | 1 | 0 | 0
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 0 | 0
Renal/Genitourinary-Other Specify (Renal and urinary disorders) | 1 | 0 | 0
Secondary malig-poss related to ca txt (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 1 | 0
Syncope (fainting) (Nervous system disorders) | 1 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT00712582/Prot_SAP_000.pdf